CLINICAL TRIAL: NCT01497717
Title: Efficacy of Humira in Behcet Patients With Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Dr. Yolanda Braun, Senior Rheumatologist, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0488-09RMB; A06-197 (Other: Protocol Number of Collaborator - Abbott Company)
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Arthritis; Behcet
MeSH Terms: conditions — Arthritis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab, Behcet with arthritis (Experimental)
  Interventions: Drug: Adalimumab (Humira)

INTERVENTIONS:
Drug: Adalimumab (Humira) — Open label pilot trial.
  The study includes 3 phases :
  1. Open label treatment period of 24 weeks.
  2. Extension follow -up (3 years): Patients who responded well to study drug and their disease relapsed within the first 12 weeks following study drug interruption will be eligible to receive the study drug for 3 years in order to comply with the Israeli Ministry of Health requirements.
  3. Safety follow-up: For patients who withdraw from either the open label treatment period or extension period, for another 24 weeks.
  Other Names: Anti TNF monoclonal antibodies

SUMMARY:
Hypothesis - Behcet's disease is a multisystemic chronic relapsing inflammatory disease, classified among the vasculitides. The clinical manifestations include mucocutaneous lesions, articular, ocular, vascular, gastrointestinal and/or central nervous system involvement.

The aetiology of Behcet's disease is unknown, however. Experimental evidence suggests that TNF-α may play an important role in the pathogenesis of the disease.

To date, case reports and small open-short term studies report the efficacy of anti-TNFα therapy (Infliximab and Etanercept), especially regarding ocular and mucocutaneous involvement in Behcet.

There are no double blind long term studies on larger number of patients regarding the efficacy of anti-TNFα, especially Humira in healing arthritis +/- other manifestations of the disease.

DETAILED DESCRIPTION:
Study Design (including visit schedule, dosing and procedures/methods):

Screen visit, 1st visit -treatment initiation, follow-up visits - after 1 month and afterwards every 8 weeks for 24 weeks.

Screen visit: informed consent, medical history,inclusion and exclusion criteria, pregnancy test, vital signs, physical examination, joint evaluation (no. of tender joints, no. of swollen joints), patient/investigator global disease activity, pain VAS, HAQ, Behcet Disease Current Activity Forms (BDACF), ECG, PPD and chest X-ray screening for tuberculosis, routine labs (performed at local HMO as a routine follow-up of the patient treatment with DMARD's): CBC, blood chemistry, ESR, CRP, urinalysis, HbsAg and AntiHCV, immunology labs (rheumatoid factor, anti-CCP, anti nuclear antibody - ANA).

An induration of greater than 5 mm will be considered a positive PPD reaction.

Follow up visits .: Vital signs, joint evaluation, patient/investigator global disease activity, pain VAS, HAQ, BDACF, routine labs (performed at local HMO as a routine follow-up of the patient treatment with DMARD's): CBC, blood chemistry, ESR, CRP, urinalysis, research blood samples for storage.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent and comply with the requirements of the study protocol.
2. Patients with Behcet disease ,who fulfilled the International Study group criteria for Behcet Disease.
3. Experienced an inadequate response to previous or current treatment with one or more DMARDs because of inadequate efficacy or side effects.
4. DMARDS and/or corticosteroids (< or equivalent to 10mg/d prednisone) permitted if stable for at least 4 weeks prior to screening. NSAIDs permitted if stable for at least 2 weeks prior to screening.
5. Active peripheral arthritis at screening (tenderness and swelling of at least 3 small joints or one large joint) OR axial involvement (active enthesitis or spondylitis)
6. Age 18-80 years.
7. If female and of childbearing potential, a negative urine pregnancy test within 2 weeks prior to therapy, and using reliable means of contraception.

Exclusion Criteria:

1. Rheumatic autoimmune disease other than Behcet (Rheumatoid arthritis, SLE, scleroderma, etc).
2. Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders.
3. Known active bacterial, viral, fungal, mycobacterial or other infection, or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
4. History of lymphoproliferative or hematologic malignancy. History of any other type of cancer in the past 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction in DAS28 | Week 24
  The proportion of patients with improvement in arthritis (DAS 28) at week 24 -changes from screening in DAS 28 , HAQ, , CRP. ANOVA analysis and descriptive statistics. An interim evaluation of the above parameters will be performed at week 16 (visit 4) and yearly afterwards for 3 more years in those patients who will continue drug study during the extension period

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Braun, MD, Principal Investigator — Rheumatology Unit, Rambam Health Care Campus, B. Rappaport Faculty of Medicine, Technion - Institute of Technology, Israel
Locations (1):
- Rheumatology Unit, Rambam Health Care Campus, Haifa, Israel